CLINICAL TRIAL: NCT01498185
Title: A Randomized, Double-Blind, Placebo-controlled, Parallel Group, Phase 2 Trial to Explore the Safety, Pharmacokinetics and Pharmacodynamics of Dapagliflozin as an Add-on to Insulin Therapy in Subjects With Type 1 Diabetes Mellitus
Brief Title: BMS - Safety, Pharmacokinetics (PK) and Pharmacodynamics (PD) of Dapagliflozin in Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Astra Zeneca, Bristol-Myers Squibb (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB102-072
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1: Dapagliflozin (1 mg) (Experimental)
  Interventions: Drug: Dapagliflozin
- Arm 2: Dapagliflozin (2.5 mg) (Experimental)
  Interventions: Drug: Dapagliflozin
- Arm 3: Dapagliflozin (5 mg) (Experimental)
  Interventions: Drug: Dapagliflozin
- Arm 4: Dapagliflozin (10 mg) (Experimental)
  Interventions: Drug: Dapagliflozin
- Arm 5: Placebo matching Dapagliflozin (Experimental)
  Interventions: Drug: Placebo matching Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 1 mg, Once daily, 14 days
  Arms: Arm 1: Dapagliflozin (1 mg); Arm 2: Dapagliflozin (2.5 mg); Arm 3: Dapagliflozin (5 mg); Arm 4: Dapagliflozin (10 mg)
Drug: Placebo matching Dapagliflozin — Tablets, Oral, 0 mg, Once daily, 14 days
  Arms: Arm 5: Placebo matching Dapagliflozin

SUMMARY:
To obtain safety and tolerability information in patients with type 1 diabetes where Dapagliflozin is added on to Insulin (for 14 days)

DETAILED DESCRIPTION:
Study Classification : Safety, Pharmacokinetics and Pharmacodynamics

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes with central lab Glycosylated hemoglobin (A1C) ≥ 7.0% and ≤ 10.0%
* Insulin use for at least 12 months and initiation immediately after diagnosis of diabetes
* Method of Insulin administration [multiple daily injections (MDI) or continuous subcutaneous Insulin infusion (CSII)] stable ≥ 3 months
* Stable basal Insulin dose ≥ 2 weeks
* Ages 18 to 65 years
* Central laboratory C-peptide value of < 0.7 ng/mL
* Body mass index (BMI) 18.5 to 35.0 kg/m2

Exclusion Criteria:

* History of type 2 diabetes mellitus (T2DM), maturity onset diabetes of young (MODY), pancreatic surgery or chronic pancreatitis
* Oral hypoglycemic agents
* History of diabetes ketoacidosis (DKA) within 24 weeks
* History of hospital admission for glycemic control within 6 months
* Frequent episodes of hypoglycemia (2 unexplained within 3 months) or hypoglycemic unawareness
* Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) or Serum total bilirubin > 2X Upper limit of normal (ULN)
* Abnormal Free T4 [if screening Thyroid Stimulating Hormone (TSH) abnormal]
* Estimated glomerular filtration rate (eGFR) Modification of Diet in Renal Disease (MDRD) formula ≤ 60 mL/min/1.73m2
* Cardiovascular (CV)/Vascular Diseases within 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- United States (12):
  - Profil Institute For Clinical Research, Inc., Chula Vista, California
  - Va San Diego Healthcare System, San Diego, California
  - La Biomed Research Inst. At Harbor Ucla Med Ctr., Torrance, California
  - Compass Research Phase 1, Llc, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Vince And Associates Clinical Research, Overland Park, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Jasper Clinic, Inc., Kalamazoo, Michigan
  - Kansas City University Of Medicine And Biosciences, Kansas City, Missouri
  - Regional Medical Clinic-Endocrinology, Rapid City, South Dakota
  - Dallas Diabetes & Endocrine Center, Dallas, Texas

REFERENCES:
- [Derived] Melin J, Tang W, Rekic D, Hamren B, Penland RC, Boulton DW, Parkinson J. Dapagliflozin Pharmacokinetics Is Similar in Adults With Type 1 and Type 2 Diabetes Mellitus. J Clin Pharmacol. 2022 Oct;62(10):1227-1235. doi: 10.1002/jcph.2062. Epub 2022 May 2. PMID 35403243
- [Derived] Henry RR, Rosenstock J, Edelman S, Mudaliar S, Chalamandaris AG, Kasichayanula S, Bogle A, Iqbal N, List J, Griffen SC. Exploring the potential of the SGLT2 inhibitor dapagliflozin in type 1 diabetes: a randomized, double-blind, placebo-controlled pilot study. Diabetes Care. 2015 Mar;38(3):412-9. doi: 10.2337/dc13-2955. Epub 2014 Sep 30. PMID 25271207
- See also: MB102072_Clinical_Study_Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3117&filename=MB102072_Clinical_Study_Protocol_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 171 participants enrolled, 76 completed a screening period. Of these 76 participants, 70 were randomized and received treatment. Of these 70 participants, 62 completed double-blind treatment period.
Groups:
- Placebo + Insulin; Dapagliflozin 1 mg + Insulin; Dapagliflozin 2.5 mg + Insulin; Dapagliflozin 5 mg + Insulin; Dapagliflozin 10 mg + Insulin: Tablets, oral, once daily for 2 weeks
Period: Overall Study
Arm/Group | Placebo + Insulin | Dapagliflozin 1 mg + Insulin | Dapagliflozin 2.5 mg + Insulin | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin
Started | 13 | 13 | 15 | 14 | 15
Completed | 12 | 12 | 15 | 11 | 12
Not Completed | 1 | 1 | 0 | 3 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2 | 1
Not completed — No longer met criteria, etc | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Insulin | Dapagliflozin 1 mg + Insulin | Dapagliflozin 2.5 mg + Insulin | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin | Total
Number analyzed (Participants) | 13 | 13 | 15 | 14 | 15 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.5 (12.18) | 33.7 (9.11) | 35.7 (13.93) | 34.8 (14.00) | 37.5 (15.24) | 35.3 (12.86)
Age, Customized [Number; unit: Participants]
  Younger than 45 years | 10 | 11 | 11 | 9 | 10 | 51
  45 years and older | 3 | 2 | 4 | 5 | 5 | 19
Sex/Gender, Customized [Number; unit: Participants]
  Male | 8 | 5 | 11 | 8 | 8 | 40
  Female | 5 | 8 | 4 | 6 | 7 | 30
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 11 | 11 | 14 | 14 | 12 | 62
  Black/African American | 1 | 1 | 1 | 0 | 2 | 5
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Other | 1 | 0 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in 7-Point Glucose Monitoring (7-PGM) at Day 7
Description: 7-PGM was measured as milligrams per deciliter (mg/dL) by a central laboratory. Baseline was defined as the assessment on Day -1, prior to the start date and time of the first dose of the double-blind study medication. 7-PGM included the average of all available glucose values before and 2-hour (hr) after each meal (breakfast, lunch, dinner) as well as bedtime. Measurements were on Day -1, and Day 7 in the double-blind period.
Time Frame: From Baseline to Day 7
Population: All randomized participants who received study medication and had nonmissing values at baseline and Day 7
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo + Insulin | Dapagliflozin 1 mg + Insulin | Dapagliflozin 2.5 mg + Insulin | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin
Number analyzed (Participants) | 13 | 12 | 12 | 14 | 12
mg/dL | -16.52 (14.6316) | -19.01 (10.9920) | -17.29 (7.1451) | -23.40 (9.4334) | -17.55 (10.8430)
Statistical Analysis 1: Comparison: Placebo + Insulin vs Dapagliflozin 1 mg + Insulin; Test type: Superiority or Other; Descriptive statistics — No formal statistical testing was performed to compare between treatment groups; Mean Difference (Final Values) = -2.50, 95% CI 2-sided [-40.85 to 35.86], Standard Error of Mean 18.5425
Statistical Analysis 2: Comparison: Placebo + Insulin vs Dapagliflozin 2.5 mg + Insulin; Test type: Superiority or Other; Descriptive statistics — No formal statistical testing was performed to compare between treatment groups; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-35.36 to 33.82], Standard Error of Mean 16.7228
Statistical Analysis 3: Comparison: Placebo + Insulin vs Dapagliflozin 5 mg + Insulin; Test type: Superiority or Other; Descriptive statistics — No formal statistical testing was performed to compare between treatment groups; Mean Difference (Final Values) = -6.88, 95% CI 2-sided [-42.21 to 28.45], Standard Error of Mean 17.1548
Statistical Analysis 4: Comparison: Placebo + Insulin vs Dapagliflozin 10 mg + Insulin; Test type: Superiority or Other; Descriptive statistics — No formal statistical testing was performed to compare between treatment groups; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-39.22 to 37.16], Standard Error of Mean 18.4617

2. Secondary Outcome: Dapagliflozin Pharmacokinetic Parameters on Day 7 - Maximum Observed Plasma Concentration (Cmax)
Description: Serial blood samples were collected predose 0 hr, and hr 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 in the double-blind period. Individual subject PK parameter values were derived by non-compartmental methods by a validated PK analysis program, Kinetica®. Actual sampling times were used for PK calculations and nominal times were used for generation of mean plasma concentration-time plots and summaries. Pre-dose sample collection times were changed from negative numbers (based on elapsed time to dose) to zero for the purpose of calculating PK parameters. The Cmax was recorded directly from experimental observations.
Time Frame: Day 7 (0 hr to 24 hr post dose)
Population: Randomized subjects who took at least one dose of dapagliflozin with adequate pharmacokinetic parameter profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dapagliflozin 1 mg + Insulin | Dapagliflozin 2.5 mg + Insulin | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin
Number analyzed (Participants) | 12 | 14 | 14 | 13
ng/mL | 12.18 (45.93) | 24.19 (32.46) | 66.11 (41.07) | 134.34 (29.33)

3. Secondary Outcome: Dapagliflozin Pharmacokinetic Parameters on Day 7 - Time of Maximum Observed Plasma Concentration (Tmax)
Description: Serial blood samples were collected predose 0 hr, and hr 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 in the double-blind period. Individual subject PK parameter values were derived by non-compartmental methods by a validated PK analysis program, Kinetica®. Actual sampling times were used for PK calculations and nominal times were used for generation of mean plasma concentration-time plots and summaries. Pre-dose sample collection times were changed from negative numbers (based on elapsed time to dose) to zero for the purpose of calculating PK parameters. The Tmax was recorded directly from experimental observations.
Time Frame: Day 7 (0 hr to 24 hr post dose)
Population: Randomized subjects who took at least one dose of dapagliflozin with adequate pharmacokinetic parameter profiles
Measure: Mean (Full Range); unit: hour
Arm/Group | Dapagliflozin 1 mg + Insulin | Dapagliflozin 2.5 mg + Insulin | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin
Number analyzed (Participants) | 12 | 14 | 14 | 13
hour | 1.04 (45.93) [0.4 to 4.0] | 1.08 (32.46) [0.2 to 3.0] | 1.03 (41.07) [0.5 to 4.0] | 1.27 (29.33) [0.0 to 4.0]

4. Secondary Outcome: Dapagliflozin Pharmacokinetic Parameters on Day 7 - Area Under the Concentration-Time Curve in One Dosing Interval (AUC[TAU])
Description: Serial blood samples were collected predose 0 hr, and hr 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 in the double-blind period. Individual subject PK parameter values were derived by non-compartmental methods by a validated PK analysis program, Kinetica®. Actual sampling times were used for PK calculations and nominal times were used for generation of mean plasma concentration-time plots and summaries. Pre-dose sample collection times were changed from negative numbers (based on elapsed time to dose) to zero for the purpose of calculating PK parameters. The concentrations below the lower limit of quantitation (<LLOQ) were set as "missing" for the calculation of PK parameters as well as summary statistics. AUC[TAU], was calculated by a mixture of logand linear-trapezoidal summations.
Time Frame: Day 7 (0 hr to 24 hr post dose)
Population: Randomized subjects who took at least one dose of dapagliflozin with adequate pharmacokinetic parameter profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dapagliflozin 1 mg + Insulin | Dapagliflozin 2.5 mg + Insulin | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin
Number analyzed (Participants) | 12 | 14 | 14 | 13
ng*h/mL | 48.42 (23.71) | 127.17 (32.30) | 269.09 (27.25) | 600.01 (48.33)

5. Secondary Outcome: Dapagliflozin 3-O-glucuronide Pharmacokinetic Parameters on Day 7 - Maximum Observed Plasma Concentration (Cmax)
Description: as for outcome 2
Time Frame: Day 7 (0 hr to 24 hr post dose)
Population: Randomized subjects who took at least one dose of dapagliflozin with adequate pharmacokinetic parameter profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dapagliflozin 1 mg + Insulin | Dapagliflozin 2.5 mg + Insulin | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin
Number analyzed (Participants) | 12 | 14 | 14 | 13
ng/mL | 10.58 (31.73) | 21.96 (44.48) | 49.22 (43.33) | 106.68 (26.80)

6. Secondary Outcome: Dapagliflozin 3-O-glucuronide Pharmacokinetic Parameters on Day 7 - Time of Maximum Observed Plasma Concentration (Tmax)
Description: as for outcome 3
Time Frame: Day 7 (0 hr to 24 hr post dose)
Population: Randomized subjects who took at least one dose of dapagliflozin with adequate pharmacokinetic parameter profiles
Measure: Mean (Full Range); unit: hour
Arm/Group | Dapagliflozin 1 mg + Insulin | Dapagliflozin 2.5 mg + Insulin | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin
Number analyzed (Participants) | 12 | 14 | 14 | 13
hour | 1.42 (45.93) [0.9 to 4.0] | 1.83 (32.46) [1.0 to 4.0] | 1.57 (41.07) [0.8 to 4.0] | 1.84 (29.33) [0.5 to 6.0]

7. Secondary Outcome: Dapagliflozin 3-O-glucuronide Pharmacokinetic Parameters on Day 7 - Area Under the Concentration-Time Curve in One Dosing Interval (AUC[TAU])
Description: as for outcome 4
Time Frame: Day 7 (0 hr to 24 hr post dose)
Population: Randomized subjects who took at least one dose of dapagliflozin with adequate pharmacokinetic parameter profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dapagliflozin 1 mg + Insulin | Dapagliflozin 2.5 mg + Insulin | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin
Number analyzed (Participants) | 12 | 14 | 14 | 13
ng*h/mL | 49.63 (29.85) | 132.38 (36.06) | 262.58 (33.33) | 567.77 (39.59)

8. Secondary Outcome: Pharmacokinetic Parameters on Day 7 - Ratio of Metabolite (RM) to Parent AUC[TAU]
Description: Serial blood samples were collected predose 0 hr, and hr 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 in the double-blind period. Individual subject PK parameter values were derived by non-compartmental methods by a validated PK analysis program, Kinetica®. Actual sampling times were used for PK calculations and nominal times were used for generation of mean plasma concentration-time plots and summaries. Pre-dose sample collection times were changed from negative numbers (based on elapsed time to dose) to zero for the purpose of calculating PK parameters. The concentrations below the lower limit of quantitation (<LLOQ) were set as "missing" for the calculation of PK parameters as well as summary statistics. MR was calculated as the ratio of metabolite to parent AUC(TAU), corrected for molecular weights of dapagliflozin and dapagliflozin 3-O-glucuronide (408.82 and 584.99, respectively).
Time Frame: Day 7 (0 hr to 24 hr post dose)
Population: Randomized subjects who took at least one dose of dapagliflozin with adequate pharmacokinetic parameter profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h/mL):(ng*h/mL)
Arm/Group | Dapagliflozin 1 mg + Insulin | Dapagliflozin 2.5 mg + Insulin | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin
Number analyzed (Participants) | 12 | 14 | 14 | 13
(ng*h/mL):(ng*h/mL) | 0.72 (29.29) | 0.73 (33.22) | 0.68 (25.69) | 0.66 (32.37)

ADVERSE EVENTS:
Time Frame: Onset on or after the first date of double-blind treatment and on or prior to the last day of double-blind treatment 24 weeks plus 4 days for non-serious adverse event; plus 30 days for serious adverse event.
Arm/Group | Placebo + Insulin | Dapagliflozin 1 mg + Insulin | Dapagliflozin 2.5 mg + Insulin | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/15 | 1/14 | 0/15
Other Adverse Events (participants affected / at risk) | 8/13 | 5/13 | 7/15 | 7/14 | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Insulin (N=13) | Dapagliflozin 1 mg + Insulin (N=13) | Dapagliflozin 2.5 mg + Insulin (N=15) | Dapagliflozin 5 mg + Insulin (N=14) | Dapagliflozin 10 mg + Insulin (N=15)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Insulin (N=13) | Dapagliflozin 1 mg + Insulin (N=13) | Dapagliflozin 2.5 mg + Insulin (N=15) | Dapagliflozin 5 mg + Insulin (N=14) | Dapagliflozin 10 mg + Insulin (N=15)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CATHETER SITE PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BED BUG INFESTATION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VAGINAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MICTURITION URGENCY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE IRRITATION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VITREOUS FLOATERS (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (3) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABNORMAL DREAMS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
DYSMENORRHOEA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No